CLINICAL TRIAL: NCT04853381
Title: Comparison of the Effects of Different Medical Nutrition Treatments on Symptoms and Quality of Life of Patients With Irritable Bowel Syndrome and the Acceptability Status of These Dietary Treatments by Patients
Brief Title: Comparison of the Effects of Different Nutrition Treatments on Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Nezihe Otay Lule, Research assistant, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: nolule
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: low FODMAP; gluten free diet; irritable bowel syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Diet, Gluten-Free

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1st Group: Traditional diet recommendations (Experimental): Traditional diet recommendations will apply for 4 weeks.
  Interventions: Other: dietary treatment (Traditional diet recommendations)
- 2nd Group: Low FODMAP diet (Experimental): Low FODMAP diet recommendations will apply for 4 weeks. When individuals are first enrolled in the study, they will be trained by the dietician for one hour before the medical nutrition treatment they will apply for 4 weeks.
  Interventions: Other: dietary treatment (low FODMAP)
- 3rd Group: Gluten-free diet (Experimental): Gluten-free diet recommendations will apply for 4 weeks. When individuals are first enrolled in the study, they will be trained by the dietician for one hour before the medical nutrition treatment they will apply for 4 weeks.
  Interventions: Other: dietary treatment (gluten free)
- 4th Group: Low-FODMAP gluten-free diet (Experimental): Low-FODMAP gluten-free diet recommendations will apply for 4 weeks. When individuals are first enrolled in the study, they will be trained by the dietician for one hour before the medical nutrition treatment they will apply for 4 weeks.
  Interventions: Other: dietary treatment (low FODMAP+gluten free)

INTERVENTIONS:
Other: dietary treatment (low FODMAP) — The aim of the study will be explained to the patients and the dietary treatment that will be recommended if they participate in the study will be told that they should be followed for 4 weeks. In addition, it will be notified that surveys will be conducted at the beginning and end of the 4-week period.
  Arms: 2nd Group: Low FODMAP diet
Other: dietary treatment (gluten free) — The aim of the study will be explained to the patients and the dietary treatment that will be recommended if they participate in the study will be told that they should be followed for 4 weeks. In addition, it will be notified that surveys will be conducted at the beginning and end of the 4-week period.
  Arms: 3rd Group: Gluten-free diet
Other: dietary treatment (low FODMAP+gluten free) — The aim of the study will be explained to the patients and the dietary treatment that will be recommended if they participate in the study will be told that they should be followed for 4 weeks. In addition, it will be notified that surveys will be conducted at the beginning and end of the 4-week period.
  Arms: 4th Group: Low-FODMAP gluten-free diet
Other: dietary treatment (Traditional diet recommendations) — The aim of the study will be explained to the patients and the dietary treatment that will be recommended if they participate in the study will be told that they should be followed for 4 weeks. In addition, it will be notified that surveys will be conducted at the beginning and end of the 4-week period.
  Arms: 1st Group: Traditional diet recommendations

SUMMARY:
Irritable Bowel Syndrome (IBS) is a disease associated with changes in bowel habits characterized by unexplained abdominal discomfort or pain. Common symptoms of the disease include gas, bloating, diarrhea, constipation, and common gastrointestinal problems associated with psychosocial problems. IBS makes it difficult for patients to attend school and work, reduce productivity, increase healthcare costs and negatively affect quality of life. Although IBS is not a life-threatening disease, it is a condition that must be tackled throughout life. The disease is clinically managed through dietary interventions and appropriate lifestyle changes, and pharmacological symptom-targeted or psychological treatments.

The aim of this study is to determine the effects of different dietary treatment methods on patients 'severity symptom score and quality of life, and the patients' compliance with different dietary treatments.

DETAILED DESCRIPTION:
Patients between the ages of 19-65 who applied to Gaziantep University Faculty of Medicine, Department of Gastroenterology and diagnosed with Irritable Bowel Syndrome by the physician according to the Rome IV criteria will be included in the study. The aim of the study will be explained to the patients and the dietary treatment that will be recommended if they participate in the study will be told that they should be followed for 4 weeks. In addition, it will be notified that surveys will be conducted at the beginning and end of the 4-week period. Written consent will be obtained from individuals who agree to participate in the study.

The minimum number of individuals in each group was determined to be 13 when the power was calculated as 80 at a 95% confidence interval. Individuals who accepted to participate in the study will be randomized into 4 different groups by minimization method according to age, gender, irritable bowel syndrome subtypes (diarrhea, constipation, mixed / undefined) and initial irritable bowel syndrome severity scores (mild, moderate, severe):. 1st Group: Traditional diet recommendations, 2nd Group: Low FODMAP diet, 3rd Group: Gluten-free diet, 4th Group: Low-FODMAP gluten-free diet. When individuals are first enrolled in the study, they will be trained by the dietician for one hour before the medical nutrition treatment they will apply for 4 weeks.

"Irritable Bowel Syndrome Severity Scoring Scale", "Bristol Stool Scale", "Irritable Bowel Syndrome Quality of Life Scale", "Food Consumption Frequency Survey including FODMAP Intake" and "Food Consumption Frequency Survey Including Gluten Intake" will be applied to individuals at the beginning of the study and at the end of the 4th week.

ELIGIBILITY:
Inclusion Criteria:

1. Applying to Gaziantep University Faculty of Medicine Department of Gastroenterology,
2. Between the ages of 19-65,
3. Diagnosed with Irritable Bowel Syndrome by a physician according to Rome IV criteria,
4. Patients who voluntarily accept to participate in the study will be included in the study after explaining the purpose and method of the study.

Exclusion Criteria:

1. Those with gastrointestinal organic diseases (celiac, lactose intolerance, inflammatory bowel diseases),
2. Those diagnosed with clinically important systemic diseases (diabetes, cancer, hypertension, thyroid and other endocrine system diseases),
3. Individuals diagnosed with multiple sclerosis and Parkinson's disease,
4. Individuals with established food allergies,
5. Individuals with major psychiatric diseases,
6. Individuals with eating disorders according to DSM-V criteria,
7. Individuals who have undergone major abdominal surgery,
8. Individuals who were pregnant at the time of the study will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome Severity Scoring Scale (IBS-SSS) | at baseline
  this test evaluates the severity of the disease. The overall score of IBS-SSS ranges from 0 to 500. According to this standardized survey, 75-175 points: mild symptom 175--300 points: moderate symptom > 300 points: considered to be severe symptoms.
Irritable Bowel Syndrome Severity Scoring Scale (IBS-SSS) | end of the 4th week.
  this test evaluates the severity of the disease. The overall score of IBS-SSS ranges from 0 to 500. According to this standardized survey, 75-175 points: mild symptom 175--300 points: moderate symptom > 300 points: considered to be severe symptoms.
Irritable Bowel Syndrome Quality of Life Scale (IBS-QQL) | at baseline
  This test determines the quality of life of patients with irritable bowel syndrome. Irritable Bowel Syndrome Quality of Life Scale consists of 34 items and 8 subgroups; Each item in a Likert-type scale has 5 answer options. "1 Nothing", "2 A Little"; "3 Middle"; One of the "4 Too Much" and "5 Too Much" options should be selected. According to these options, the first option is 5; The fifth option is given 1 point and the total score is calculated.
  Minimum 34 points and maximum 170 points are obtained as total points. An increase in the total score obtained from the scale indicates an increase in the quality of life associated with the disease.
Irritable Bowel Syndrome Quality of Life Scale (IBS-QQL) | end of the 4th week
  This test determines the quality of life of patients with irritable bowel syndrome. Irritable Bowel Syndrome Quality of Life Scale consists of 34 items and 8 subgroups; Each item in a Likert-type scale has 5 answer options. "1 Nothing", "2 A Little"; "3 Middle"; One of the "4 Too Much" and "5 Too Much" options should be selected. According to these options, the first option is 5; The fifth option is given 1 point and the total score is calculated.
  Minimum 34 points and maximum 170 points are obtained as total points. An increase in the total score obtained from the scale indicates an increase in the quality of life associated with the disease.
Bristol Stool Scale | at baseline
  This test questions the shape and consistency of stool in patients with irritable bowel syndrome.
  This scale aims to estimate the stool form from 7 different stool shapes. It is understood that there is improvement in the stool form as you approach the number 4 form.
Bristol Stool Scale | end of the 4th week
  This test questions the shape and consistency of stool in patients with irritable bowel syndrome.
  This scale aims to estimate the stool form from 7 different stool shapes. It is understood that there is improvement in the stool form as you approach the number 4 form.

SECONDARY OUTCOMES:
Food Consumption Frequency Survey including FODMAP Intake | at baseline
  determines the frequency of patients consuming foods containing FODMAPs.
Food Consumption Frequency Survey including FODMAP Intake | end of the 4th week
  determines the frequency of patients consuming foods containing FODMAPs.
Food Consumption Frequency Survey Including Gluten Intake | at baseline
  determines the frequency of patients consuming foods containing gluten.
Food Consumption Frequency Survey Including Gluten Intake | end of the 4th week
  determines the frequency of patients consuming foods containing gluten.

CONTACTS AND LOCATIONS:
Overall Officials: S.Mine YURTTAGUL, Study Director — Hasan Kalyoncu University
Locations (1):
- Gaziantep University, Gaziantep, Sehitkamil, Turkey (Türkiye)